CLINICAL TRIAL: NCT07314450
Title: Procedural Sedation and Analgesia for Treatment of Adults With Fractures and Dislocations in the Emergency Department
Acronym: PAINEX
Status: Recruiting | Type: Observational
Sponsor: Region Zealand (Other)
Collaborators: Zealand University Hospital (Other); Odense University Hospital (Other); Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Sophie Sværke, Principal Investigator, Region Zealand
Other Study IDs: p-2025-19278; S-20252000-95 (Other: The Committees on Health Research Ethics)
Record Dates: First submitted 2025-12-05; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pain, Procedural; Analgesia; Extremity Injury; Patient Satisfaction; Satisfaction, Personal; Satisfaction; Upper Extremity Injury; Lower Extremity Fracture; Upper Extremity Fracture; Extremity Injuries Lower
Keywords: Emergency Department; Procedural sedation and analgesia
MeSH Terms: conditions — Pain, Procedural; Agnosia; Patient Satisfaction; Personal Satisfaction; Arm Injuries; Leg Injuries; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extremity injuries: Each department will collect data on the treatment patients with the upper and lower extremity injuries receive during reduction or stabilizing treatment (procedural sedation and/or analgesia, or no treatment).
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: Usual Care — No intervention: Patients will receive usual care

SUMMARY:
The goal of this observational study is to evaluate the effectiveness and safety of different procedural sedation and analgesia methods used for adults with painful fractures requiring reduction treatment in the emergency department.

The main questions it aims to answer are:

* Which sedation and analgesia methods provide the best patient satisfaction and pain relief?
* How do different treatment methods affect clinician satisfaction and the occurrence of adverse events?

The investigators will compare different types of procedural sedative and analgesic treatments (such as systemic sedation/analgesia and regional techniques like nerve or hematoma blocks) to see which approach offers the best patient satisfaction and most effective pain control.

Participants will:

Be adult patients with upper or lower extremity fractures or joint dislocations requiring painful reduction procedures.

Receive one of the routinely used sedation or analgesia treatments (or no analgesia) during their emergency department care.

Report their pain levels and satisfaction before, during, and after treatment. Be monitored for any side effects, complications, or use of antidotes. Data will be collected over a six-month period at Odense University Hospital, Holbæk Hospital, and Zealand University Hospital, Køge, following the STROBE guidelines for observational studies.

DETAILED DESCRIPTION:
Please refer to the full protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.
2. Patients with the following injuries are eligible:

   1. Reduction treatment of shoulder dislocation
   2. Reduction treatment of elbow dislocation
   3. Reduction treatment of distal radius fractures, application of cast
   4. Reduction treatment of finger fractures/dislocation
   5. Casting treatment of upper extremity fractures

      * Proximal humerus fracture, application of fixed sling
      * Humeral shaft fracture, application of Sarmiento brace
      * Supracondylar fracture, application of angled cast
   6. Reduction treatment of hip dislocation
   7. Reduction treatment of patella dislocation
   8. Reduction of tibial shaft fracture, application of cast
   9. Reduction treatment of ankle fractures including distal tibia fracture
   10. Reduction treatment for toe fractures/dislocation
   11. Casting treatment of lower extremity fractures

       * Distal femur fracture, application of cast/traction
       * Proximal tibia fracture, application of cast or hinged brace
       * Ankle fracture, application of walker

Exclusion Criteria:

1. Unable to give informed consent (e.g. unconscious, psychotic or dementia)
2. Unwilling to participate in the study
3. Prior inclusion in the study
4. Already included in another clinical study at the same day/hospital visit
5. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients with upper and lower extremity injuries that require painful stabilizing treatment in the emergency department.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction via Numerical Rating Scale | Immediately after the procedure
  Patient satisfaction with the procedural sedation regimen will be assessed using the 11-point Numerical Rating Scale, which ranges from 0 to 10, where 0 indicates complete dissatisfaction and 10 indicates complete satisfaction. Higher scores will reflect a better outcome.
  Patients will be assessed clinically for alertness and readiness to respond before being asked the outcome questions. Only once they are awake and able to provide informed responses will the assessments be performed.

SECONDARY OUTCOMES:
Re-call of maximum pain intensity | Immediately after the procedure
  Re-call of the maximum pain intensity during the treatment procedure will be assessed using the Numerical Rating Scale, which ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Higher scores will reflect a worse outcome.
  Patients will be assessed clinically for alertness and readiness to respond before being asked the outcome questions. Only once they are awake and able to provide informed responses will the assessments be performed.
Patient satisfaction via Short Assessment of Patient Satisfaction | Immediately after the procedure
  Patient satisfaction with the sedation regimen and treatment will be assessed using the Short Assessment of Patient Satisfaction, which consists of 7 items, each scored from 0 to 4, yielding a total score ranging from 0 to 28, with the overall score reflecting a continuum from very dissatisfied to very satisfied. Higher scores will indicate greater patient satisfaction.
  Patients will be assessed clinically for alertness and readiness to respond before being asked the outcome questions. Only once they are awake and able to provide informed responses will the assessments be performed.
Clinician satisfaction with analgosedation regimen | Immediately after the procedure
  Clinician satisfaction with the analgosedation regimen will be assessed using the Numerical Rating Scale, which ranges from 0 to 10, where 0 indicates complete dissatisfaction and 10 indicates complete satisfaction. Higher scores will reflect a better outcome.
  Patients will be assessed clinically for alertness and readiness to respond before being asked the outcome questions. Only once they are awake and able to provide informed responses will the assessments be performed.
Incidence of adverse events | During and immediately after the procedure
  Incidence of the following adverse events will be recorded: hypoxia, hypotension, treatment-requiring bradycardia, nausea, vomiting, hallucinations, and the need for reversal agents (antidote medication). Each event will be reported as a dichotomous outcome (present or absent).
  Patients will be assessed clinically for alertness and readiness to respond before being asked the outcome questions. Only once they are awake and able to provide informed responses will the assessments be performed.

OTHER OUTCOMES:
Patient satisfaction via 5-point Likert Scale | Immediately after the procedure
  Patient satisfaction with the sedation regimen and treatment will be assessed using a 5-point Likert Scale, which ranges from 1 to 5, where 1 indicates very dissatisfied and 5 indicates very satisfied. Higher scores will reflect a better outcome.
  Patients will be assessed clinically for alertness and readiness to respond before being asked the outcome questions. Only once they are awake and able to provide informed responses will the assessments be performed.
Incidence of procedural amnesia | Immediately after the procedure
  Incidence of procedural amnesia will be assessed as a patient-reported outcome. Each case will be recorded as present or absent. Higher incidence reflects a better outcome.
  Patients will be assessed clinically for alertness and readiness to respond before being asked the outcome questions. Only once they are awake and able to provide informed responses will the assessments be performed.
Incidence of dissociative experience during treatment | Immediately after the procedure
  Incidence of dissociative experience during the treatment procedure will be assessed as a patient- and physician-reported outcome. Each case will be recorded as present or absent and categorized as a good or bad experience. A higher incidence of bad experiences will reflect a worse outcome, whereas a higher incidence of good experiences will reflect a better outcome.
  Patients will be assessed clinically for alertness and readiness to respond before being asked the outcome questions. Only once they are awake and able to provide informed responses will the assessments be performed.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Emergency Department, Holbæk Hospital, Holbæk, Region Sjælland
  - Emergency Department, Zealand University Hospital, Køge, Region Sjælland
  - Emergency Department, Odense University Hospital, Odense, Region Syddanmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT07314450/Prot_SAP_000.pdf